CLINICAL TRIAL: NCT02642107
Title: The Multicenter Randomized Phase 3 Trial of Individualized Elective Neck Irradiation Based on MRI in Patients With Nasopharyngeal Carcinoma
Brief Title: Individualized Elective Neck Irradiation Based on MRI in NPC Patients
Acronym: NPC-CTVn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Guilin Medical College (Other)
Responsible Party: Principal Investigator, Ling-Long Tang, associated professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5010-2015-05
Record Dates: First submitted 2015-12-16; First posted 2015-12-30 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; elective neck irradiation; upper neck irradiation; whole neck irradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elective neck irradiation (Experimental): Whole neck irradiation is given in the involved neck. Elective neck irradiation of Level II,III and Va lymph node area is given in the uninvolved neck, and Level IV and Vb lymph node area were not irradiated in the uninvolved neck.
  Interventions: Radiation: Elective neck irradiation
- Whole neck irradiation (Active Comparator): Whole neck irradiation is given regardless of the involved or uninvolved neck.
  Interventions: Radiation: Whole neck irradiation

INTERVENTIONS:
Radiation: Elective neck irradiation — Whole neck irradiation is given in the involved neck. Elective neck irradiation of Level II,III and Va lymph node area is given in the uninvolved neck, and Level IV and Vb lymph node area were not irradiated in the uninvolved neck.
  Arms: Elective neck irradiation
Radiation: Whole neck irradiation — Whole neck irradiation is given regardless of the involved or uninvolved neck.
  Arms: Whole neck irradiation

SUMMARY:
Currently, most protocols of nasopharyngeal carcinoma (NPC) of various research bodies such as the Radiation Therapy Oncology Group require routine elective irradiation to the retropharyngeal area and to levels II-V lymph nodal areas regardless of the status of nodal metastasis. Previous studies had confirmed that the pattern of cervical lymph node (LN) metastasis in NPC followed an orderly manner. Retropharyngeal LNs were the most commonly involved, followed by upper neck levels II, III, or VA nodes, and finally to the lower neck nodes including level IV and VB nodes; and the incidence of LN skip metastasis is rare, ranging from 0.5% to 7.9%. It was rare for NPC patients without neck LN metastases to experience neck failure after elective irradiation to levels II, III and VA. It was also confirmed that with unilateral LN metastases of higher-level LNs usually spread down ipsilateral LNs. Thus, the investigators conduct the non-inferior randomized trial to determine the value of elective neck irradiation in NPC patients with unilateral or bilateral uninvolved neck.

DETAILED DESCRIPTION:
Currently, most protocols of nasopharyngeal carcinoma (NPC) of various research bodies such as the Radiation Therapy Oncology Group require routine elective irradiation to the retropharyngeal area and to levels II-V lymph nodal areas regardless of the status of nodal metastasis. Previous studies had confirmed that the pattern of cervical lymph node (LN) metastasis in NPC followed an orderly manner. Retropharyngeal LNs were the most commonly involved, followed by upper neck levels II, III, or VA nodes, and finally to the lower neck nodes including level IV and VB nodes; and the incidence of LN skip metastasis is rare, ranging from 0.5% to 7.9%. It was rare for NPC patients without neck LN metastases to experience neck failure after elective irradiation to levels II, III and VA. It was also confirmed that with unilateral LN metastases of higher-level LNs usually spread down ipsilateral LNs. Thus, the investigators conduct the non-inferior randomized trial to determine the value of elective neck irradiation in NPC patients with unilateral or bilateral uninvolved neck.

ELIGIBILITY:
The eligibility criteria are: newly diagnosed, untreated, non-distant metastatic, and non-keratinizing NPC; with unilateral or bilateral uninvolved neck; aged between 18 and 65 years; Karnofsky performance-status score > 70; adequate haematological function, with a leucocyte count > 4 × 109/L, haemoglobin > 90 g/L, and a thrombocyte count > 100×109/L.

The exclusion criteria include: previous chemotherapy treatment, surgery (except diagnostic) or radiotherapy to the neck or nasopharyngeal regions; previous malignancy; lactation or pregnancy; or severe coexisting illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Regional relapse-free survival | 3 year
  The regional relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to the date of nodal relapse or death from any cause, whichever occurred first. Their differences will be compared between treatment arms using the log-rank test.

SECONDARY OUTCOMES:
Radiation-related toxicity | Within 1 month after radiotherapy for acute toxicity; long term for late toxicity
  Acute and late toxicity will be documented according to RTOG/EORTC System and the CTCAE(Common Terminology Criteria for Adverse Events). Toxicity will be summarized using descriptive statistics.
Overall survival | 3 year
  The overall survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Local relapse-free survival | 3 year
  The local relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to documented local relapse or death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Distant metastasis-free survival | 3 year
  The distant metastasis-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to documented distant metastasis or death from any cause. Their differences will be compared between treatment arms using the log-rank test.
Patient's quality-of-life: global health status | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on global health status suggest better health.
Patient's quality-of-life: physical functioning | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the functioning scales suggest better function.
Patient's quality-of-life: role functioning | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the functioning scales suggest better function.
Patient's quality-of-life: emotional functioning | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the functioning scales suggest better function.
Patient's quality-of-life: cognitive functioning | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the functioning scales suggest better function.
Patient's quality-of-life: social functioning | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the functioning scales suggest better function.
Patient's quality-of-life: fatigue | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: nausea and vomiting | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: pain | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: dyspnoea | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: insomnia | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: appetite loss | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: constipation | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: diarrhoea | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: financial difficulties | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Core 30 items (QLQ-C30) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: pain | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: swallowing | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: sense problems | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: speech problems | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: trouble social eating | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: trouble social contact | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: less sexuality | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: teeth | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: open mouth | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: dry mouth | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: sticky saliva | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: coughing | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: felt ill | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: pain killers | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: nutrition supplement | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: feeding tube | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: weight loss | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.
Patient's quality-of-life: weight gain | 3 year
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires will be used to assess quality-of-life. All items pointing to this domain are averaged and then transformed to a scale of 0-100 according to the EORTC scoring manual. Higher scores on the symptom scales indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Linglong Tang, M.D.,PhD, Principal Investigator — Sun sat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CL, Zhang N, Jiang W, Xie FY, Pei XQ, Huang SH, Wang XY, Mao YP, Li KP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Zhou GQ, Ma J, Sun Y, Chen L, Tang LL. Reduced-Volume Irradiation of Uninvolved Neck in Patients With Nasopharyngeal Cancer: Updated Results From an Open-Label, Noninferiority, Multicenter, Randomized Phase III Trial. J Clin Oncol. 2024 Jun 10;42(17):2021-2025. doi: 10.1200/JCO.23.02086. Epub 2024 Mar 20. PMID 38507662
- [Derived] Tang LL, Huang CL, Zhang N, Jiang W, Wu YS, Huang SH, Mao YP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Sun Y, Xie FY, Chen L, Zhou GQ, Ma J. Elective upper-neck versus whole-neck irradiation of the uninvolved neck in patients with nasopharyngeal carcinoma: an open-label, non-inferiority, multicentre, randomised phase 3 trial. Lancet Oncol. 2022 Apr;23(4):479-490. doi: 10.1016/S1470-2045(22)00058-4. Epub 2022 Feb 28. PMID 35240053